CLINICAL TRIAL: NCT06772220
Title: Pilot Study of Open Label Homocysteine Management Therapy in Levodopa-treated Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Joseph Quinn, OHSU Parkinson Center Director, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 25171; PF-CER-979199 (Other Grant/Funding Number: Parkinson's Foundation)
Record Dates: First submitted 2025-01-02; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Parkinson&Amp;#39;s Disease
Keywords: Parkinson's disease; Parkinson disease; homocysteine
MeSH Terms: conditions — Parkinson Disease | interventions — Folic Acid; Vitamin B 6; Vitamin B 12

STUDY DESIGN:
Intervention Model Description: Study participants with elevated homocysteine levels at the first study visit will take B vitamins for 3 months, and then have a follow-up visit. Study participants with normal homocysteine levels at the first study visit will not take the B vitamins, and will also have a follow-up visit 3 months later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B vitamin regimen (Experimental): Daily doses of 1mg folic acid, 25mg vitamin B6, and 1,000 ug vitamin B12.
  Interventions: Dietary Supplement: Folic Acid 1 MG; Dietary Supplement: Vitamin B6 25 MG; Dietary Supplement: Vitamin B12
- No vitamins (No Intervention): No vitamin intervention.

INTERVENTIONS:
Dietary Supplement: Folic Acid 1 MG — Folic Acid 1mg per day
  Arms: B vitamin regimen
Dietary Supplement: Vitamin B6 25 MG — Vitamin B6, 25mg per day
  Arms: B vitamin regimen
Dietary Supplement: Vitamin B12 — Vitamin B12, 1,000 ug per day
  Arms: B vitamin regimen

SUMMARY:
This is a research study investigating elevated homocysteine in the blood of patients with Parkinson's disease who are currently receiving treatment with levodopa. We are evaluating if elevated homocysteine can be corrected using open label B vitamin therapy, as well as the impact of homocysteine levels on cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of probable Parkinson's Disease according to Movement Disorders Society criteria.
2. Currently treated with levodopa at a minimum dose of 300 mg/day
3. Montreal Cognitive Assessment (MOCA) ≥15
4. Demonstrated capacity to provide informed consent.
5. 40-90 years of age
6. Estimated glomerular filtration rate ≥60
7. Absence of uncontrolled hypertension in medical history
8. Absence of insulin use

Exclusion Criteria:

-

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hyperhomocysteinemia and B vitamin deficiency | baseline measurement
  Plasma vitamin B12 in subjects with vs without hyperhomocysteinemia
Hyperhomocysteinemia and B vitamin deficiency | baseline measurement
  Plasma folic acid in subjects with vs without hyperhomocysteinemia
Hyperhomocysteinemia and B vitamin deficiency | baseline measurement
  Plasma pyridoxine in subjects with vs without hyperhomocysteinemia

SECONDARY OUTCOMES:
Hyperhomocysteinemia and cognitive assessments | From enrollment to the end of treatment at 3 months
  Change in total Braincheck score in subjects with vs without hyperhomocysteinemia
Hyperhomocysteinemia and measurement of neurofilament light in plasma | From enrollment to the end of treatment at 3 months
  Change in plasma neurofilament level in subjects with vs without hyperhomocysteinemia

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Quinn, MD, Principal Investigator — Oregon Health & Science University (OHSU)
Locations (1):
- Oregon Health & Science University (OHSU), Portland, Oregon, United States